CLINICAL TRIAL: NCT02986932
Title: A Study to Evaluate the Safety and Feasibility of Blood-Brain Barrier (BBB) Opening Using Transcranial MR-Guided Focused Ultrasound With Intravenous Ultrasound Contrast Agents in Patients With Early Alzheimer's Disease
Brief Title: Blood-Brain-Barrier Opening Using Focused Ultrasound With IV Contrast Agents in Patients With Early Alzheimer's Disease
Acronym: BBB-Alzheimers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL001
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Alzheimer Disease
Keywords: Blood-Brain Barrier
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Transcranial ExAblate
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BBB opening (Experimental): ExAblate focused ultrasound under MRI-guidance delivered through the intact human skull in conjunction with timed intravenous ultrasound contrast agents (Definity®) to temporarily and focally open the BBB.
  Interventions: Device: BBB opening

INTERVENTIONS:
Device: BBB opening — Open BBB using ExAblate focused ultrasound and (Definity®) contrast agent

SUMMARY:
This is a prospective, non-randomized, single-arm, feasibility study to evaluate the safety and initial effectiveness of opening of the Blood-Brain Barrier with intravenous contrast agents using the ExAblate Neuro System in patients with early stage Alzheimer's Disease.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, non-randomized, feasibility, phase I trial to evaluate the safety of focal BBB opening using the ExAblate® Transcranial (220 kHz) system and Definity® ultrasound contrast in 6 patients with mild Alzheimer's Disease. This phase I trial will be divided into two stages. In the first stage, patients will undergo small volume BBB opening, establishing the minimum required sonication parameters to open the BBB, as evidenced by gadolinium enhancement on T1-weighted MRI. Stage I is defined as a discrete region of approximately 9 mm x 9 mm area in the right frontal lobe. Multiple sonications will be performed starting at low energy and ramping up until the BBB is observed to open. The subjects will then be removed from the ExAblate® Neuro device and followed for safety for 30 days. If the subject experienced BBB opening without any serious adverse effects (such as brain edema), then the subject may proceed to Stage two where a larger volume (2.5-3.0 cm) will be targeted. Subjects will be followed for an additional 60 days for safety and preliminary effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Probable AD consistent with NIA/AA criteria (McKhann, Alzheimer & Dementia 2011)
2. Modified Hachinski Ischemia Scale (MHIS) score of <= 4.
3. Mini Mental State Exam (MMSE) scores 18-28
4. Short form Geriatric Depression Scale (GDS) score of <= 6
5. Has a Florbetaben PET scan consistent with the presence of amyloid pathology in the proposed target region (right frontal lobe)
6. Able to communicate sensations during the ExAblate® MRgFUS procedure.

Exclusion Criteria:

1. MRI findings:

   * Active infection/inflammation
   * Acute or chronic hemorrhages, specifically > 4 lobar microbleeds, and no siderosis or macrohemorrhages
   * Tumor/space occupying lesion
   * Meningeal enhancement
2. More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp
3. Clips or other metallic implanted objects in the skull or the brain, except shunts; other metallic objects implanted in body
4. Significant cardiac disease or unstable hemodynamic status including:
5. Uncontrolled hypertension on medication or abnormal ECG
6. Medications known to increase risk of hemorrhage, (e.g.: patients should be off of aspirin or another anticoagulants for at least 7 days prior to treatment) or anticoagulants (class I and III) or off Avastin for 30 days
7. History of a bleeding disorder, coagulopathy or a history of spontaneous hemorrhage or use of anticoagulants
8. Abnormal coagulation profile (PLT < 100,00/μl), PT (>14 sec) or PTT (>36 sec), and INR > 1.3
9. No more than 1 non-strategic lacune <1.5 cm
10. Known cerebral or systemic vasculopathy
11. Significant depression and at potential risk of suicide
12. Known sensitivity/allergy to gadolinium (an alternative product may be used), Definity or any of its components.
13. Any contraindications to MRI scanning such as metallic implants, claustrophibia or too large for MRI scanner
14. Untreated, uncontrolled sleep apnea
15. Impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2
16. Does not have a reliable caregiver in frequent contact with the patient and can accompany the patient to the clinic and treatment or be available by telephone at designated times. Participants living in retirement homes may be included. Caregiver not willing to sign the Informed Consent Form
17. Respiratory: chronic pulmonary disorders e.g. severe emphysema, pulmonary vasculitis, or other causes of reduced pulmonary vascular cross-sectional area, patients with a history of drug allergies, asthma or hay fever, and multiple allergies where the benefit/risk of administering Definity® is considered unfavorable by the study physicians in relation to the product monograph for Definity.
18. Currently in a clinical teial involving investigational product.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in contrast enhancement (intensity) following BBB disruption | Immediately post treatment
  Change in contrast enhancement (intensity) following BBB disruption to pre-sonication images as a comparative ratio measured in percent as read from MR images and normalized to the contralateral hemisphere

SECONDARY OUTCOMES:
Change in amyloid uptake | 30 days after treatments
  Change in amyloid uptake as compared to pre treatment scans in the targeted region
Adverse events | 90 days
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
MMSE - Mini Mental State Examination | 30 days
  Treatment effect on patients' dementia state
ADAS-Cog - Alzheimer's Disease Assessment Scale - Cognitive Behavior subscales | 30 days
  Treatment effect on patients' Alzheimer's disease symptoms
NPI - Neuropsychiatry Inventory | 30 days
  Treatment effect on patients' dementia
GDS - Geriatric Depression Scale | 30 days
  Treatment effect on patients' depression
ADCS-ADL - Alzheimer's Disease Co-operative Study - Activities of Daily Living Inventory | 30 days
  Treatment effect on patients' activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Nir Lipsman, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mathew AS, Gorick CM, Price RJ. Multiple regression analysis of a comprehensive transcriptomic data assembly elucidates mechanically- and biochemically-driven responses to focused ultrasound blood-brain barrier disruption. Theranostics. 2021 Oct 11;11(20):9847-9858. doi: 10.7150/thno.65064. eCollection 2021. PMID 34815790